CLINICAL TRIAL: NCT04510233
Title: Ivermectin Inhalation Forms in the Management of COVID-19 Egyptian Patients
Brief Title: Ivermectin Nasal Spray for COVID19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kamal Mohammed Okasha, Vice President, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IvrInh
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ivermectin nasal spray (Experimental): Ivermectin administered as nasal spray (one ml in each nostril two times daily)
  Interventions: Drug: Ivermectin nasal
- Ivermectin oral (Experimental): Ivermectin administered orally (one tablet 6 mg three times daily) for 72 hours plus the standard care of COVID-19 cases.
  Interventions: Drug: Ivermectin oral
- standard care (Experimental): COVID-19 cases will receive standard of care [oxygen via masks or ventilators]
  Interventions: Other: standard care

INTERVENTIONS:
Drug: Ivermectin nasal — Ivermectin nasal spray one ml in each nostril two times daily
  Other Names: ivermectin
  Arms: Ivermectin nasal spray
Drug: Ivermectin oral — Ivermectin oral (one tablet 6 mg three times daily)
  Other Names: ivermectin
  Arms: Ivermectin oral
Other: standard care — oxygen via masks or ventilators
  Arms: standard care

SUMMARY:
The global escalation of COVID19 pandemic has put the health care system under pressure with urgent need for treatment. In the absence of vaccine and approved drug against SARS-COV2 over the past 6 months, the health authorities were obliged to re-purpose existing drugs to fight this pandemic.

DETAILED DESCRIPTION:
Ivermectin is a well-known FDA-approved pan antiparasitic drug with high safety profile and potential therapeutic effects against COVID 19. It has been previously investigated as an antiviral agent. It showed 5000 fold reduction of SARS COV 2 viral RNA in-vitro studies.

However, some researchers questioned its efficacy in the oral form as very high doses will be required to achieve a proper tissue concentration and viricidal effect in the respiratory system.

Our hypothesis is that, since COVID-19 has shown to be particularly damaging to the respiratory system, using inhaled forms of Ivermectin will deliver the drug directly to the infection site and make it a treatment option.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate severity who are confirmed to be positive for SARS COV 2.

Exclusion Criteria:

* patients with severe form of COVID-19 or those who are on ventilatory support or those with cytokine storm

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PCR of SARS-Cov2 RNA | 14 days
  Negative PCR result of SARS-Cov2 RNA in COVID19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Okasha, PhD, Principal Investigator — Tanta Univesity faculty of Medicine

IPD SHARING:
Plan to Share IPD: No